CLINICAL TRIAL: NCT03924375
Title: Serum Pepsinogen After Helicobacter Pylori Eradication for the Gastric Cancer Prevention
Brief Title: Serum Pepsinogen After H. Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2019
Record Dates: First submitted 2019-04-20; First posted 2019-04-23 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Helicobacter Pylori Eradication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biospecimen would be obtained for urease test (commercial name: CLOtest).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori has been recognized as a major pathogen in gastric carcinogenesis. Current guidelines recommend the H. pylori "test-and-treat" strategy for the purpose of primary and secondary gastric cancer prevention. Considering the "point of no return" theory, however, H. pylori eradication cannot reduce the risk of gastric cancer in subjects with gastric atrophy and intestinal metaplasia. The intragastric hypoacidic environment is associated with the risk of intestinal-type gastric cancer development. Recently, the secretory ability of the stomach can be measured using the serum pepsinogen (PG) assay.

DETAILED DESCRIPTION:
This study aimed to evaluate the change of serum PGs after H. pylori eradication success and identify the optimal timing of eradication.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* Serologic markers including serum pepsinogen can be measured

Exclusion Criteria:

* Age < 20 or > 70 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected subjects who underwent an upper gastrointestinal endoscopy were enrolled in this study at a single, tertiary-care, academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Serum pepsinogen change after H. pylori eradication | after 8 weeks
  Serum pepsinogen recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Jun-Hyung, M.D., Principal Investigator — Digestive Disease Center, Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No